CLINICAL TRIAL: NCT06831552
Title: A Randomized Phase II Trial Evaluation of the Addition of the Resource Intervention to Support Equity (RISE) to Usual Supportive Care for Children With Newly Diagnosed High-Risk Neuroblastoma
Brief Title: Resource Intervention to Support Equity (RISE) in High-Risk Neuroblastoma
Acronym: RISE in HR NBL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Kira Bona, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-600
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Neuroblastoma; High-risk Neuroblastoma
Keywords: Neuroblastoma; High-risk Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: RISE Intervention + Usual Supportive Care (Experimental): Participants will be randomized in a 1:1 ratio and stratified according to treatment group and Household Material Hardship (HMH) severity score. Participant parents/guardians will complete:
  * Orientation visit in-person, by phone, or virtually with survey
  * Access to usual supportive oncology care comprised of social workers, resource specialists and/or psychosocial oncology teams
  * Meeting with a benefits counselor by phone or virtually and follow up meetings if needed
  * Fixed amount of cash assistance 2x monthly
  * 3 months survey
  * 6 month survey
  Interventions: Behavioral: RISE Intervention
- Arm 2: Usual Supportive Care (No Intervention): Participants will be randomized in a 1:1 ratio and stratified according to treatment group and HMH severity score. Participant parents/guardians will complete:
  * Orientation visit in-person, by phone, or virtually with survey
  * Access to usual supportive oncology care comprised of social workers, resource specialists and/or psychosocial oncology teams
  * 3 month survey
  * 6 month survey

INTERVENTIONS:
Behavioral: RISE Intervention — Income-poverty targeted, supportive care intervention that includes direct cash transfers delivered by the Fund for Guaranteed Income, a non-profit organization, along with benefits counseling to discuss the risk of means-tested benefits loss or reduction. Funds will be dispersed to families via debit card or through personal banking, PayPal, or Venmo on a twice monthly basis for a total of twelve disbursements (6-months). Meetings with a benefits counselor will be conducted by the HIPAA-compliant video conference platform, Zoom.
  Other Names: Pediatric Resource Intervention to Support Equity
  Arms: Arm 1: RISE Intervention + Usual Supportive Care

SUMMARY:
The goal of this study is to test if the addition of a novel income-poverty targeted supportive care intervention (Pediatric Resource Intervention to Support Equity [Pediatric RISE]) to usual supportive care for low-income children with high-risk neuroblastoma can improve parent- and child-centered outcomes.

Participants will be randomized to receive one of the following for 6-months:

* Usual supportive care alone or
* Usual supportive care plus Pediatric RISE

DETAILED DESCRIPTION:
This is a randomized Phase II trial evaluating the addition of the RISE supportive care equity intervention to usual supportive care for poverty-exposed children participants with newly diagnosed high-risk neuroblastoma. Participants will be randomized into one of two groups: Usual supportive care or Pediatric RISE plus usual supportive care. Randomization means a participant is placed into a study group by chance.

The research study procedures include screening for eligibility, in-person or virtual appointments, and surveys.

Participation in this research study is expected to last for about 6-months.

It is expected that about 84 participants will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

Patient cohort: The randomized Phase II multi-center RISE intervention will be conducted among a population of poverty-exposed children with high-risk neuroblastoma. Poverty will be a priori defined as parent-reported low-income (<200% Federal Poverty Level). Children receiving treatment for cancer at study sites will serve as the study cohort, with parents/guardians as survey informants and intervention recipients on behalf of their minor children given that parents (not children) typically manage household finances.

* Patient newly diagnosed with high-risk neuroblastoma
* Patient has established care at study site and initiated cancer-directed therapy
* Patient has not yet initiated Induction Cycle 3
* Patient aged 0-17 years at the time of consent
* Parent/guardian screened positive for self-reported low-income (<200% Federal Poverty) *
* Family primary residence in MA, PA, IL, CA, WA, CT, GA, WI and OH
* Both patients co-enrolled on ANBL2131 or those receiving standard of care therapy at their center are eligible to participate
* Patients of all languages are eligible to participate

Exclusion Criteria:

* Foreign national family receiving care as an Embassy-pay patient.
* Child or household member receiving SSI

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Household Material Hardship (HMH) Score Reduction Rate | Baseline (T1) and 6-months (end-intervention; T3)
  HMH score reduction rate is defined as the proportion of patients achieving at least 1 domain reduction in (food, housing, utility or transportation insecurity). HMH scores range from 0 to 4, with scores of 0 indicating no hardship (unexposed) and scores of 1-4 indicating the presence of hardship (exposed). Patients who are unexposed to HMH at baseline (HMH score of 0) are excluded from the analysis.

SECONDARY OUTCOMES:
Pediatric-Modified Comprehensive Score for Financial Toxicity (COST) | 3-months (end-of-induction; T2) and 6-months (end-intervention; T3)
  Financial toxicity will be assessed with the 12-item modified COST measure. Each item is rated on a 0-4 scale, yielding a total score range of 0-48, with higher scores indicating better financial well-being. The final COST score will be calculated per established methods. A change of approximately 5 points is considered a minimally important difference (MID), representing a clinically meaningful change in financial toxicity.
Parent Psychological Distress (Kessler-6) Score Change from Baseline to 6 Months | Baseline (T1) and 6-months (end-intervention; T3)
  Psychological distress will be assessed using the 6-item Kessler-6 scale. The scale includes 6 items scored from 0 ('none of the time') to 4 ('all of the time'), yielding a total score ranging from 0 to 24, with higher scores indicating greater psychological distress. A reduction in scores of approximately 2.8 points is considered a minimally important difference (MID), representing a clinically meaningful improvement in psychological distress.
Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Abilities Score Change from Baseline to 6 Months | Baseline (T1) and 6-months (end-intervention; T3)
  The PROMIS Applied Cognition-Abilities short form is an 8-item measure assessing subjective learning and memory, attention and concentration, executive function, and processing speed. Responses are scored on a scale of 1-5, and the total score is converted to a T-score with a mean of 50 and a standard deviation (SD) fixed at 10. Higher scores suggest better perceived cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Kira Bona, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Dr. Kira Bona. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication